CLINICAL TRIAL: NCT01129258
Title: A Phase 1 Placebo-Controlled Trial to Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Multiple Escalating Oral Doses of PF-04991532 in Adult Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Multiple Dose Study of PF-04991532 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B2611004
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders
Keywords: phase 1; safety and tolerability; pharmacokinetics; PK; pharmacodynamics; PD; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04991532 (Experimental)
  Interventions: Drug: PF-04991532
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04991532 — Subjects will be dosed wtih PF-04991532 for 14 days. The tentative dosing schedule is 30, 100, 300, 1000, and 1500 mg QD, and 150 and 500 mg BID). Doses shown may be adjusted upwards or downwards and may be adjusted to include intermediate doses. All doses will be administered as tablets (10, 50, and 150 mg strengths). In each cohort 9 subjects will receive PF-04991532 and 3 will receive placebo.
  Arms: PF-04991532
Drug: Placebo — Placebo to match PF-04991532 will be provided. Subjects will be dosed for 14 days. In each cohort 9 subjects will receive PF-04991532 and 3 will receive placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of PF-04991532 following multiple (14 days) escalating oral doses in patient wtih type 2 diabetes.

DETAILED DESCRIPTION:
Safety/Tolerability, PK, and PD

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus who are taking metformin only. Treatment should be stable, where this is defined as no change in the treatment, including dose, over the past 2 months. Subjects treated with a sulfonylurea (SU) or a dipeptidyl peptidase-4 inhibitor (DPP-4i) in combination with metformin may be eligible if washed off the SU or DPP-4i to metformin only for a minimum of 4 weeks before dosing. Subjects being switched over from an SU and metformin or a DPP-4i and metformin to metformin only will still need to meet the fasting glucose requirements on Day -2 as defined in the protocol.
* Body Mass Index (BMI) of 18.5 to 45.0 kg/m2; and a total body weight >50 kg (110 lbs).
* Fasting C-peptide >0.8 ng/mL.
* HbA1c >/=7% and >/=10%. If the patient requires to be washed off an SU or DPP-4i, the HbA1c limits will be >/=6.5% and </=9%.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease. Subjects who have chronic conditions other than T2DM (for example, hypercholesterolemia or hypertension) but are controlled by either diet or stable (for the last 2 months) doses of medications may be included as well.
* Evidence or history of diabetic complications with significant end-organ damage.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* History of stroke, transient ischemic attack, or myocardial infarction within the past 6 months.
* History of coronary artery bypass graft or stent implantation.
* Clinically significant peripheral vascular disease.
* Any history or clinical evidence of congestive heart failure, NYHA Classes II-IV.
* Current history of angina/unstable angina.
* ECG findings suggestive of asymptomatic myocardial ischemia or QTc >470 msec at screening.
* One or more self-reported episodes of hypoglycemia within the last 3 months, or two or more self-reported episodes of hypoglycemia within the last 6 months.
* Screening or Day -2 fasting (>/=8 hours) glucose, </=90 or >/=270 mg/dL, confirmed by a single repeat if deemed necessary.
* A positive urine drug screen.
* Use of tobacco or nicotine-containing products in excess of the equivalent of 10 cigarettes per day.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Certain concomitant medications are excluded, as defined in the protocol.
* Screening supine blood pressure >/=160 mm Hg (systolic) or >/=100 mm Hg (diastolic).
* Certain laboratory values (for example, triglyceride and liver function test results).
* Pregnant or nursing females; females of childbearing potential.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety Endpoints: Safety and tolerability of PF-04991532 will be assessed by physical examinations, adverse event monitoring, 12-lead ECGs, vital sign, and clinical safety laboratory measurements. | 5 months
Single-Dose PK Endpoints for PF-04991352: Cmax, Tmax, and AUC(0-tau). | 5 months
Multiple-Dose PK Endpoints for PF-04991532: Cmax(ss), Tmax(ss), AUC(0-tau,ss), AUC(0-last), half-life, Cmin(ss), Cav(ss), Ae%, CL/F, Vz/F, CLrenal; accumulation ratios AUC(0-tau,ss)/AUC(0-tau,sd) and Cmax(ss)/Cmax(sd), as the data permit. | 5 months
PD Endpoint: glucose excursion (change from Day -1 baseline) in response to a liquid meal test (MMTT) on Days 1 and 14. | 5 months

SECONDARY OUTCOMES:
Insulin and C-peptide (changes from Day -1 baseline) during an MMTT on Days 1 and 14. | 5 months
Mean daily glucose (change from Day -1 baseline) on Days 1 and 14. | 5 months
Fasting plasma glucose (change from Day -1 baseline) on Days 1, 3, 6, 10, and 14. | 5 months
Lipids (change from Day -1 baseline), including: TG, TC, HDL-cholesterol, LDL-cholesterol, FFA, beta-OHB, and ACAC, at times specified in the SOA. | 5 months
Lactate (change from Day -1 baseline), at times specified in the SOA. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611004&StudyName=Multiple%20Dose%20Study%20of%20PF-04991532%20in%20Patients%20with%20Type%202%20Diabetes